CLINICAL TRIAL: NCT05730816
Title: MAGIC-AKI: Magnesium for the Prevention of Hyperthermic Intraoperative Cisplatin-Associated AKI
Brief Title: MAGIC AKI: Magnesium for the Prevention of HIOC-Associated AKI
Acronym: MAGIC-AKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shruti Gupta, Director of Onconephrology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023p000276; K23DK125672 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; Magnesium Sulfate; intraoperative cisplatin
MeSH Terms: conditions — Mesothelioma | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Sulfate (Experimental): The IV Mg will start at 1 g/hour (25 ml/hour) within one hour following induction of anesthesia and stabilization of the patient. The infusion will continue for 24 hours and serum Mg levels will be monitored every 4 hours (+/-1 hour) for 28 hours following initiation of the Mg. Dose adjustments to the Mg infusion will be made as necessary to reach target serum Mg levels (3-5 mg/dl).
  Interventions: Drug: Magnesium sulfate
- Normal Saline (Placebo Comparator): Patients randomized to placebo will receive an equal volume of normal saline (0.9% NS) placebo which will be administered as a continuous infusion at 25 ml/hour. The infusion will continue for 24 hours.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium sulfate — Intravenous infusion of magnesium sulfate prior to intraoperative chemotherapy with cisplatin.
  Arms: Magnesium Sulfate
Drug: Normal Saline — Intravenous infusion of normal saline.
  Arms: Normal Saline

SUMMARY:
In this research study, investigators will test whether prophylactic high-dose IV Mg administration attenuates the risk of AKI in patients with malignant mesothelioma receiving intraoperative chemotherapy (HIOC) with cisplatin compared to placebo

.

DETAILED DESCRIPTION:
In this phase 2, open-label randomized, placebo-controlled trial, investigators will test whether prophylactic high-dose IV Mg administration attenuates the risk of HIOC-associated AKI in patients with malignant mesothelioma undergoing surgery with HIOCC. Investigators will randomly assign 130 patients to receive IV Mg versus an equal volume of normal saline (0.9% NS) placebo, of whom it is anticipated 80 will complete the study. Investigators will also collect blood and urine pre- and postoperatively for exploration of secondary outcomes.

Investigators will screen for eligibility at participant's preoperative visit with their thoracic surgeon. Intravenous magnesium will be administered as a continuous infusion, soon after induction and stabilization by anesthesia in the operating room. The magnesium drip will start at 1 g/hour and will be titrated to achieve target levels of 3-5 mg/dl. The total duration of the infusion will be 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. • Adult patients (≥18 years old) with malignant mesothelioma undergoing surgery with HIOC with Dr. Raphael Bueno or another BWH thoracic surgeon

Exclusion Criteria:

1. eGFR<45 ml/min/1.73m2 on either screening labs or preoperative labs, or end-stage kidney disease receiving renal replacement therapy. Screening labs refer to those obtained at the preoperative visit with the surgeon or within 90 days prior, whereas preoperative labs are obtained on the day of admission (typically one to three days priors to surgery).
2. Serum Mg >3 mg/dl on either screening labs or preoperative labs
3. Pregnant/breastfeeding
4. Neuromuscular disease (e.g., myasthenia gravis, amyotrophic lateral sclerosis, multiple sclerosis, muscular dystrophy, myositis)
5. Coronary artery disease, defined as any of the following in the prior year: a positive stress test; coronary angiogram indicating 1 or more vessels with >70% stenosis; percutaneous coronary intervention with stents; or coronary artery bypass graft surgery
6. Sinus bradycardia, defined as a heart rate (HR) <55 beats per minute (bpm) detected on any ECG in the preceding 6 months
7. High grade AV block (2nd degree AV block type II or 3rd degree AV block) without a pacemaker
8. Positive COVID test in the 10 days prior to surgery
9. Prisoner
10. Hypersensitivity to Mg sulfate
11. Concurrent participation in a study with an alternative experimental therapy that may interact with IV Mg
12. Any condition that, in the view of the PI, might place the patient at increased risk or compromise the integrity of the study
13. Conflict with other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-04-03 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
AUC of SCr measured daily over 7 days in Mg- versus placebo-treated patients | 7 days
  The primary endpoint is the area under the curve (AUC) of SCr measured daily over 7 days in Mg- versus placebo-treated patients
Composite Global Rank | 7 days
  As a secondary endpoint, investigators will construct a composite global rank endpoint in which the highest rank is assigned to those who die within 7 days, the second highest rank is assigned to those who survive but require RRT within 7 days, and all others ranked according to their SCr AUC, since RRT and death are important competing risks.

SECONDARY OUTCOMES:
Incident AKI | 7 days
  Urine output <0.5 ml/kg/h x consecutive 6 hours in the first 48 hours following surgery with HIOC (this will only be assessed for the first 48 hours, as patients are transferred out of the ICU and/or their foley is removed, which prevents accurate hourly assessment of UOP); An absolute increase in SCr ≥0.3 mg/dl within 48 hours; C) A relative increase in SCr ≥50% compared to the baseline value in the first 7 days; D) Receipt of RRT in the first 7 days
Composite outcome of RRT/in-hospital death | 7 days
  Composite outcome
Maximum AKI stage | 7 days
  Based on KDIGO staging
Renal tubular injury | 2 days
  AUC of uNGAL, uKIM-1, and pKIM-1 at hours +4, +12, and +36 in relation to HIOC administration
AUC for platinum concentrations | 2 days
  Using blood and urine collected at various time points
Vasoactive-inotropic score (VIS) | 2 days
  Assessed every 4 hours for the first 24 hours, and then every 8 hours for the next 24 hours, in relation to the start of the Mg infusion. The VIS is a validated method for integrating all vasoactive medications (i.e., vasopressors and inotropes) and their doses on an hourly basis into a single measure, and has been used in multiple settings
Proportion of patients with serum Mg levels in the 3-5 mg/dl range in the treatment group | 1 day
  Between hours +8 and +24 in relation to the start of the Mg infusion
New onset of atrial fibrillation | 7 days
  Confirmed on an EKG
Myocardial injury | 7 days
  Defined as clinical evidence of myocardial injury and a troponin level above the 99th percentile

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Gupta, MD, MPH, Principal Investigator — Brigham and Women's Hospital; David E. Leaf, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu